CLINICAL TRIAL: NCT01609647
Title: Comparison of Prasugrel and Clopidogrel Reloading on High Platelet Reactivity in Clopidogrel-loaded Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Reloading Prasugrel or Clopidogrel on High Platelet Reactivity Before Percutaneous Coronary Intervention
Acronym: PRAISE-HPR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, MD. Director, Regional Clinical Trial Center. Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRAISE-HPR
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Acute Coronary Syndrome
Keywords: High plate reactivity unit after loading dose of clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): Reloading with prasugrel 20mg & followed by administration of 5mg/day for 30 days
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Reloading with clopidogrel 300mg and followed by administration of clopidogrel 75 mg/day for 30 days
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Reloading with prasugrel 20mg and followed by daily administration of prasugrel 5mg for 30 days
  Other Names: Effient
  Arms: Prasugrel
Drug: Clopidogrel — Reloading with clopidogrel 300mg and followed by daily administration of clopidogrel 75mg for 30 days
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
High platelet reactivity unit (PRU) after loading dose clopidogrel in patients undergoing percutaneous coronary intervention (PCI) is related to high risk of short and long term recurrent ischemic events including stent thrombosis.

The investigators hypothesize that additional loading of prasugrel in patients with high PRU after clopidogrel loading would be superior to additional loading of clopidogrel in reducing platelet reactivity and thereby result in lower risk of short term recurrent ischemic events.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with acetylsalicyclic acid (ASA) and additional clopidogrel is now standard regimen for the prevention of recurrent ischemic events in patients who undergo PCI.

But decreased effect of clopidogrel in a group of patients was reported and they are known to be associated with high risk of recurrent ischemic event. Decreased effect of clopidogrel is mainly resulted from decreased function to metabolite prodrug, clopidogrel to active form of drug.

Prasugrel, newer thienopyridine has been recently developed and showed advantages to clopidogrel. Prasugrel is known to have shorter onset time to achieve steady state level than clopidogrel and constant pharmacologic effect regardless of patient diversity.

High PRU after loading dose clopidogrel in patients undergoing PCI is known to be related to increased risk of short and long term recurrent ischemic events including stent thrombosis. Prasugrel has been reported to be effective in reducing platelet reactivity in patients showing resistance to clopidogrel and high PRU.

The investigators hypothesize that additional loading of prasugrel in patients with high PRU after clopidogrel loading would be superior to additional loading of clopidogrel in reducing platelet reactivity and thereby result in reduced risk of short term recurrent ischemic events.

The investigators plan to include 70 acute coronary syndrome patients who are planned to undergo PCI and show high platelet reactivity. Most patients with ACS administer loading dose of ASA and clopidogrel as soon as they are assumed to be ACS.

The investigators plan to perform platelet reactivity test by VeryfyNow (VN) before PCI and enroll patients with high PRU defined by 235 or more. They are to randomly administered additional 300mg of clopidogrel or 20mg of prasugrel.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* Patients planned to undergo percutaneous transluminal coronary angioplasty
* Patients who agreed to the experimental plan which was permitted by IRB

Exclusion Criteria:

* Low body weight (<50kg)
* Urgent PCI for ACS
* Use of glycoprotein IIb/IIIa inhibitor in recent 24hrs or planned to
* History of transient ischemic attack
* History of upper gastrointestinal bleeding in recent 6 months
* Renal dysfunction defined as serum creatinine > 2.5 mg/dl
* Severe hepatic dysfunction defined as serum transaminase > 3 times normal limit
* Bleeding tendency
* Anticoagulation treatment including warfarin
* Thrombocytopenia defined by platelet < 100,000/ml
* Anemia defined by hemoglobin < 10 g/dl
* Contraindication for study drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HPR at 24 hours | 24 hours
  Persistently high platelet reactivity after PCI. PRU is measured by methods of VerifyNow device and HPRU is defined as PRU of 240 or more.

SECONDARY OUTCOMES:
MACE | 30 days (1 month)
  Major adverse cardiovascular events consist of cardiac death, myocardial infarction, stroke, stent thrombosis, cardiac enzyme (CRP, CK-MB, Troponin-I)
Bleeding | 30 days (1 month)
  Major, minor or minimal bleeding defined by TIMI(thrombolysis in myocardial infarction) bleeding criteria
HPRs | 4 hours after PCI, 30 days after PCI
  Persistently high platelet reactivity 4 hours and 30 days after PCI. PRU is measured by methods of VerifyNow device and HPRU is defined as PRU of 240 or more.
Periprocedural myocardial infarction | 48 hours after PCI
  Cardiac troponin value is >5x99th percentile upper reference plus either (1) evidence of prolonged ischaemic chest pain (>20min) or (2) ischaemic ST changes or new pathological Q waves, or (3) angiographic evidence of a side branch occlusion, slow-flow or no-reflow, embolization, or (4) imaging evidence of new regional wall motion abnormality.
Periprocedural myocardial injury | 48 hours after PCI
  Cardiac troponin (cTn) value is ≤5x99th percentile upper reference limit (URL) after PCI and cTn value was normal before the PCI or cTn value is >5x99th percentile URL in absence of ischaemic chest pain or ST changes, with normal angiographic and imaging findings.

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, Principal Investigator — Director, Regional Clinical Trial Center
Locations (1):
- DongA University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Guo LZ, Kim MH, Shin ES, Ann SH, De Jin C, Cho YR, Park JS, Park K, Park TH, Lee MS, Serebruany VL. Thienopyridine reloading in clopidogrel-loaded patients undergoing percutaneous coronary interventions: The PRAISE study. Int J Cardiol. 2016 Nov 1;222:639-644. doi: 10.1016/j.ijcard.2016.08.027. Epub 2016 Aug 4. PMID 27517654
- [Derived] Lee DH, Kim MH, Park TH, Park JS, Park K, Zhang HZ, Seo JM, Lee MS. Comparison of prasugrel and clopidogrel reloading on high platelet reactivity in clopidogrel-loaded patients undergoing percutaneous coronary intervention (PRAISE-HPR): a study protocol for a prospective randomized controlled clinical trial. Trials. 2013 Feb 28;14:62. doi: 10.1186/1745-6215-14-62. PMID 23448344